CLINICAL TRIAL: NCT04065048
Title: A Single-center Open-label Study to Determine the Effect of Diet on Microbiome Signatures in Crohn's Disease Patients
Brief Title: A Dietary Intervention Study on the Microbiome in Crohn's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University of California, Davis (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Abigail Basson, PostDoctoral Fellow, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09411; 1P30DK097948 (NIH)
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Crohn Disease
Keywords: diet; inflammatory bowel disease; gut microbiome
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: This is an open label single center study to compare the effect of a soy-based diet or an identical diet without soy on the composition and metabolite production of gut bacteria in Crohn's disease (CD) patients in remission or active disease, and in healthy controls. Crohn's subjects will be pre-screened by the treating gastroenterologist for eligibility criteria during their normally scheduled appointment. The treating gastroenterologist will ask suitable patients whether they are interested in participating in the described dietary intervention study during the patient appointment. Initial verbal consent will be obtained by the treating gastroenterologist. Healthy controls will be recruited in the same manner, as well as via a hospital flyer advertisement. Subjects will then be contacted by the study investigator to schedule a screening visit (visit 1) and if study eligibility is confirmed, and informed consent provided, enrolled into the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soy-based diet (Experimental): Participants will be randomized to follow a soy-based diet for 7 days. The diet will be preceded by a 12-hr overnight fast.
  Interventions: Other: Soy based diet
- Regular diet (Active Comparator): Participants will be randomized to follow a diet without soy for 7 days. The diet will be preceded by a 12-hr overnight fast.
  Interventions: Other: Non-soy based diet

INTERVENTIONS:
Other: Soy based diet — The diet will be based on the detailed descriptions according to the American Heart Association, US Food and Drug Administration (FDA), and the Soyfoods Association of North America Website, which all promote soy products as having beneficial nutrient profiles with a daily consumption of 25 grams or more of soy protein (average serving = 6.25 grams), upper limit of 50g.
  Arms: Soy-based diet
Other: Non-soy based diet — Diet of identical composition to the soy diet with the exception of soy.
  Arms: Regular diet

SUMMARY:
This protocol is designed to compare the effectiveness of a soy-based diet or identical diet without soy given to patients with Crohn's disease (CD) in remission, patients with active CD, or healthy controls. The assigned diet will be compared to participant 'baseline' (pre-diet) in terms of its ability to change the gut bacteria and fecal butyrate, an important short-chain fatty acid (SCFA) that limits bowel inflammation, a characteristic of this debilitating disease.

DETAILED DESCRIPTION:
The inflammatory bowel disease (IBD) subtype, Crohn's disease (CD) is a chronic and relapsing inflammatory disorder of the gastrointestinal tract. Although the precise etiology of IBD is not known, evidence suggests that environmental factors, including diet, contribute to its pathogenesis. A soy-based diet has been demonstrated to have numerous health benefits. This single-center open-label study will compare the effectiveness of a soy-based diet or an identical diet without soy to change the gut microbiota composition and fecal butyrate concentration to that of baseline (pre-diet) in patients with CD (remission or active disease) and healthy control subjects without CD. Participants will follow either a soy-based diet or an identical diet without soy to which they will be randomized for 7 days. No data collection or other study procedures will take place until the potential participant provides written informed consent to participate in the research study. The informed consent, screening, enrollment, and baseline data collection which make up visit 1 can occur on the same day or be completed across several days.

ELIGIBILITY:
Inclusion Criteria:

* CD subjects: Documented diagnosis of Crohn's disease. Control subjects: no documented diagnosis of CD.
* CD subjects: Harvey Bradshaw Index (HBI) score <4 ('CD remission'), or with HBI score >8 ('CD moderate disease')
* Capable of providing consent to participate
* Access to technology that permits the daily completion of study related activities
* Able to receive and have an adult sign for food shipments delivered to a work or home environment.
* Negative pregnancy test at screening visit in females of childbearing potential
* Able to take oral nutrition and medication intake for 3 months prior to and at time of study enrolment.
* 'CD remission' subjects: No change in 'IBD related' medications within 8 weeks prior to normally scheduled appointment with treating gastroenterologist (pre-screening): biologics, immunosuppressants, corticosteroids.

Exclusion Criteria:

* Short bowel syndrome.
* Hospitalized patients
* Body mass Index <19 kg/m or ≥35.
* Known clinically significant liver/gallbladder/pancreatic disease/dysfunction
* Individuals who lack consent capacity, including the mentally ill, prisoners, cognitively impaired participants, dementia patients.
* Uncontrolled Diabetes Type I type II
* Known drug abuse.
* Known parasitic disease of the digestive system. symptomatic intestinal stricture.
* Presence of an ostomy.
* Known concurrent malignancy.
* Other conditions that would be a contraindication to and of the study diets (e.g. Soy, peanut, wheat, gluten allergy.) or preclude the participant from completing the study
* Start of new 'IBD related' medications within 8 weeks prior to enrollment: biologics, immunosuppressants, corticosteroids.
* Documented C difficile colitis within four weeks of screening
* Well-founded doubt about the patient's cooperation.
* Existing pregnancy or lactation.
* Current participation in another diet intervention, simultaneous participation in another clinical trial, or participation in any other dietary intervention trial within the last 30 days.
* History of <3 natural bowel movements per week.
* Unable to access to technology that permits the daily completion of study related activities.
* Currently consuming a soy-based diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Cominelli, MD, PhD, Principal Investigator — Case Western Reserve University, School of Medicine, Gastroenterology
Locations (1):
- University Hospitals Digestive Health Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Study results or individual subject results such as investigational tests will not be shared with the research participants or others unless deemed medically necessary. Result of this research and management of intellectual property will adherence to the NIH Grant Policy on Sharing of Unique Research Resources including the Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources issued March 5, 2003.
  Publication of data during the project and/or at the end of the project shall be consistent with normal scientific practices. Research data which documents, supports, and validates research findings will be made available after the main findings from the final research data set have been accepted for publication.

REFERENCES:
- [Background] Wu GD, Chen J, Hoffmann C, Bittinger K, Chen YY, Keilbaugh SA, Bewtra M, Knights D, Walters WA, Knight R, Sinha R, Gilroy E, Gupta K, Baldassano R, Nessel L, Li H, Bushman FD, Lewis JD. Linking long-term dietary patterns with gut microbial enterotypes. Science. 2011 Oct 7;334(6052):105-8. doi: 10.1126/science.1208344. Epub 2011 Sep 1. PMID 21885731
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Thia K, Faubion WA Jr, Loftus EV Jr, Persson T, Persson A, Sandborn WJ. Short CDAI: development and validation of a shortened and simplified Crohn's disease activity index. Inflamm Bowel Dis. 2011 Jan;17(1):105-11. doi: 10.1002/ibd.21400. PMID 20629100

RESULTS

PARTICIPANT FLOW:
Groups:
- Crohn's on Soy Diet: Participants with Crohn's disease randomly assigned the Soy-based diet for 7 days. The diet will be preceded by a 12-hr overnight fast.
  Soy based diet: The diet will be based on the detailed descriptions according to the American Heart Association, US Food and Drug Administration (FDA), and the Soyfoods Association of North America Website, which all promote soy products as having beneficial nutrient profiles with a daily consumption of 25 grams or more of soy protein (average serving = 6.25 grams), upper limit of 50g.
- Crohn's on Non-Soy Diet: Participants with Crohn's disease randomly assigned the non-Soy diet for 7 days. The diet will be preceded by a 12-hr overnight fast.
  Non-soy based diet: Diet of identical composition to the soy diet with the exception of soy.
- Healthy Controls on Soy Diet: Healthy participants (without Crohn's disease) randomly assigned the Soy-based diet for 7 days. The diet will be preceded by a 12-hr overnight fast.
  Soy based diet: The diet will be based on the detailed descriptions according to the American Heart Association, US Food and Drug Administration (FDA), and the Soyfoods Association of North America Website, which all promote soy products as having beneficial nutrient profiles with a daily consumption of 25 grams or more of soy protein (average serving = 6.25 grams), upper limit of 50g.
- Healthy Controls on Non-Soy Diet: Healthy participants (without Crohn's disease) randomly assigned the non-Soy diet for 7 days. The diet will be preceded by a 12-hr overnight fast.
  Non-soy based diet: Diet of identical composition to the soy diet with the exception of soy.
Period: Overall Study
Arm/Group | Crohn's on Soy Diet | Crohn's on Non-Soy Diet | Healthy Controls on Soy Diet | Healthy Controls on Non-Soy Diet
Started | 18 | 17 | 16 | 16
Completed | 16 | 15 | 14 | 15
Not Completed | 2 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Crohn's on Soy Diet: Participants with Crohn's disease randomly assigned the Soy-based diet for 7 days. The diet will be preceded by a 12-hr overnight fast.
  .
- Crohn's on Non-Soy Diet: Participants with Crohn's disease randomly assigned the non-Soy diet for 7 days. The diet will be preceded by a 12-hr overnight fast.
- Healthy Controls on Soy Diet: Healthy participants (without Crohn's disease) randomly assigned the Soy-based diet for 7 days. The diet will be preceded by a 12-hr overnight fast.
- Healthy Controls on Non-Soy Diet: Healthy participants (without Crohn's disease) randomly assigned the non-Soy diet for 7 days. The diet will be preceded by a 12-hr overnight fast.
- Total: Total of all reporting groups
Arm/Group | Crohn's on Soy Diet | Crohn's on Non-Soy Diet | Healthy Controls on Soy Diet | Healthy Controls on Non-Soy Diet | Total
Number analyzed (Participants) | 16 | 15 | 14 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.43 (12.72) | 48.53 (11.30) | 36.14 (13.05) | 35.2 (14.25) | 41.55 (13.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 11 | 12 | 41
  Male | 8 | 5 | 3 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 15 | 14 | 14 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 3 | 1 | 7
  White | 13 | 15 | 9 | 11 | 48
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 14 | 15 | 60
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.15 (6.34) | 30.23 (6.46) | 28.32 (6.19) | 28.74 (5.78) | 28.93 (6.32)

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of Symptomatic Remission, Without Worsening of Any Existing Disease Activity During Study Period
Description: The primary aim will measure the Crohn's Disease Activity Index (CDAI) at the enrollment and end of study visit. CDAI scores can range from 0 to ~600 (A score of less than 150 corresponds to relative disease quiescence (remission); 150 to 219, mildly active disease; 220 to 450, moderately active disease; and greater than 450, severe disease). Herein, a cut-off value of <150 was selected so that most patients below this threshold would be rated by physicians as 'very well'. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point [i.e., value at 7 days (post) minus value at baseline/enrollment (pre)].
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Crohn's Patients on Soy Diet; Crohn's Patients on Non-soy Diet: CDAI value at 7 days minus value at baseline
Arm/Group | Crohn's Patients on Soy Diet | Crohn's Patients on Non-soy Diet
Number analyzed (Participants) | 16 | 15
score on a scale | -31.63 (57.91) | -27.57 (56.62)
Statistical Analysis 1: Comparison: Crohn's Patients on Soy Diet vs Crohn's Patients on Non-soy Diet; Test type: Other; p = 0.469, t-test, 2 sided

2. Primary Outcome: Change in Fecal Myleoperoxidase (MPO) Activity
Description: Change in fecal myleoperoxidase (MPO) activity at day 7 vs day 0.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ug/mg
Arm/Group | Crohn's on Soy Diet | Crohn's on Non-Soy Diet | Healthy Controls on Soy Diet | Healthy Controls on Non-Soy Diet
Number analyzed (Participants) | 16 | 15 | 14 | 15
ug/mg | -0.691 (1.471) | 0.7336 (1.483) | -0.0995 (0.767) | 0.5209 (1.036)
Statistical Analysis 1: Comparison: Crohn's on Soy Diet vs Crohn's on Non-Soy Diet vs Healthy Controls on Soy Diet vs Healthy Controls on Non-Soy Diet; Test type: Other; p = 0.0093, ANOVA

3. Secondary Outcome: Changes to Functional Composition of Gut Microbiota
Description: Secondary outcome will focus on changes to the functional composition of fecal gut microbiota, including bacterial butryate production after the diet intervention.
Time Frame: measured after the 7-day diet intervention
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Percentage of Subjects Who Continue Diet Following Completion of Study
Description: To assess the percentage of patients who intend to continue the study diets when prepared food is no longer provided without cost, and the reasons for discontinuation of either diet (compared to resuming usual food habits).
Time Frame: 6 months
Population: participants who responded to 6 month survey
Measure: Count of Participants; unit: Participants
Groups:
- Crohn's Participants on Soy Diet: Crohn's patients assigned a soy diet
- Crohn's Patients on Non-Soy Diet: Crohn's patients assigned a non-Soy diet
- Healthy Control Participants on Soy Diet: Healthy control participants assigned a soy diet
- Healthy Participants on Non-soy Diet: Healthy control participants assigned non-soy diet
Arm/Group | Crohn's Participants on Soy Diet | Crohn's Patients on Non-Soy Diet | Healthy Control Participants on Soy Diet | Healthy Participants on Non-soy Diet
Number analyzed (Participants) | 12 | 8 | 7 | 6
Participants | 8 | 5 | 4 | 1
Statistical Analysis 1: Comparison: Crohn's Participants on Soy Diet vs Crohn's Patients on Non-Soy Diet vs Healthy Control Participants on Soy Diet vs Healthy Participants on Non-soy Diet; Test type: Other; p = 0.2487, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 7 day diet intervention period
Groups:
- Crohn's on Soy Diet: Participants with Crohn's disease randomly assigned the Soy-based diet for 7 days.
- Crohn's on Non-Soy Diet: Participants with Crohn's disease randomly assigned the non-Soy diet for 7 days.
- Healthy Controls on Soy Diet: Healthy participants (without Crohn's disease) randomly assigned the Soy-based diet for 7 days
- Healthy Controls on Non-Soy Diet: Healthy participants (without Crohn's disease) randomly assigned the non-Soy diet for 7 days.
Arm/Group | Crohn's on Soy Diet | Crohn's on Non-Soy Diet | Healthy Controls on Soy Diet | Healthy Controls on Non-Soy Diet
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 0/15 | 1/14 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crohn's on Soy Diet (N=16) | Crohn's on Non-Soy Diet (N=15) | Healthy Controls on Soy Diet (N=14) | Healthy Controls on Non-Soy Diet (N=15)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | NA | 1 (1) | NA

LIMITATIONS AND CAVEATS:
The COVID pandemic posed a significant challenge that impeded the accrual of patients. The first participant was enrolled in 2019. However due to COVID, further participant enrollment only recommenced in 2021

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT04065048/Prot_SAP_000.pdf